CLINICAL TRIAL: NCT02933619
Title: ProMRI ICD/CRT-D Post Approval Study
Status: Completed | Type: Observational
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ProMRI PAS
Record Dates: First submitted 2016-10-10; First posted 2016-10-14 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Tachyarrhythmia
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Following product approval, confirmation of appropriate VF episode detection after MRI exposure of the ProMRI ICD/CRT-D systems and to evaluate left ventricular pacing threshold changes post-MRI.

ELIGIBILITY:
Inclusion Criteria:

* ProMRI ICD/CRT-D system enabled with BIOTRONIK Home Monitoring.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ProMRI ICD/CRT-D system enabled with BIOTRONIK Home Monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 24249 (Actual)
Dates: Start 2016-08; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Proportion of ICD/CRT-D subjects with a ≥ 5 second delay in post-MRI VF detection. | Up to 5 years post-approval
  Primary objectives will be analyzed once 25 subjects implanted with the ProMRI ICD system have been identified with a documented true VF episode post-MRI.
Proportion of LV pacing leads with a LV pacing threshold increase > 1V between pre-MRI and one-month post-MRI. | Up to 5 years post-approval

SECONDARY OUTCOMES:
Workflow compliance following MR exposure | Up to 5 years post-approval
  Proportion of subjects with appropriate restoration of tachycardia detection and ICD therapy post-MRI.
Left ventricular sensing attenuation | Up to 5 years post-approval
  Proportion of subjects who experience left ventricular sensing amplitude attenuation >50% between pre-MRI and 30 days post-MRI.